CLINICAL TRIAL: NCT06148545
Title: Efektifitas Pemberian Zat Besi Dan Vitamin D Terhadap Status Besi Pada Anak Dengan Anemia Defisiensi Besi
Brief Title: Effect of Iron and Vitamin D Supplementation to Iron Status in Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nadirah Rasyid Ridha (Other)
Collaborators: Hasanuddin University (Other)
Responsible Party: Sponsor-Investigator, Nadirah Rasyid Ridha, Paediatrician, Hasanuddin University
Organization: Hasanuddin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UH23020108
Record Dates: First submitted 2023-11-16; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Iron Deficiency, Anaemia in Children
Keywords: vitamin D; Iron status; Iron deficiency anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: children with a diagnosis of iron deficiency anemia age 1-5 years. Patients were divided into two groups, namely group A which received standard therapy (Fe preparations) 3 mg/kgBW/day, and group B (which received standard therapy combination vitamin D, 400IU).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron supplementation (Experimental): Children with a diagnosis of iron deficiency anemia. Patients who received standard therapy (Fe preparations) 3 mg/kg BW/day for 4 weeks, were then checked again for complete blood count, serum fe, and serum ferritin.
  Interventions: Drug: Elemental iron
- Iron and Vitamin D supplementation (Experimental): Children with a diagnosis of iron deficiency anemia. Patients who received standard therapy (Fe preparations) 3 mg/kgBW/day and received standard therapy combination vitamin D, 400 IU for 4 weeks, were then checked again for complete blood count, serum fe, and serum ferritin.
  Interventions: Drug: Elemental iron and Vit D

INTERVENTIONS:
Drug: Elemental iron — Group A who received standard therapy (Fe preparations) 3 mg/kg BW/day
  Other Names: Iron supplementation
  Arms: Iron supplementation
Drug: Elemental iron and Vit D — Group B received standard therapy (Fe preparations) 3 mg/kgBW/day combination with vitamin D, 400IU).
  Other Names: Iron supplementation with Vitamin D
  Arms: Iron and Vitamin D supplementation

SUMMARY:
Iron and vitamin D are two essential micronutrients for the normal growth of young children, and their deficiencies are still a major health problem in developing countries, including Indonesia. A significant association between vitamin D deficiency and anemia has been reported throughout the world. Several studies in various populations all over the world suggest a high degree of association between Iron deficiency anemia and vitamin D deficiency. It is still controversial which deficiency causes the other but this association should be addressed in view of a better treatment proposal. The aim of the present study was to determine the effect of vitamin D supplementation on iron status in iron deficiency anemia.

DETAILED DESCRIPTION:
This research is a randomized controlled trial study conducted in Makassar, South of Sulawesi, Indonesia from April to October 2023. This study was conducted on children with a diagnosis of iron deficiency anemia. Patients were divided into two groups, namely group A which received standard therapy (Fe preparations) 3 mg/kgBW/day, and group B (which received standard therapy combination vitamin D, 400IU).

The inclusion criteria in this study were children aged 1-5 years, diagnosed with iron deficiency anemia, and parents/caregivers willing to include their children in this study. Children who had received iron preparation, and previous blood transfusion were excluded in this study. Patients who refused blood tests after giving therapy for 4 weeks were declared dropouts.

Researchers will provide informed consent to parents/caregivers of children who met the research criteria. Anamnesis, general physical examination, and complete blood count (CBC) analysis were carried out: hemoglobin (Hb), Red Blood cell (RBC), Mean erythrocyte volume (MCV), Mean erythrocyte hemoglobin (MCH), Reticulocytes, serum iron, and serum ferritin. Iron deficiency anemia if the level of hemoglobin <11 g/dL, microcytic Hypochromia, serum ferritin < 30 pg/dl, then given iron and vitamin D preparation for 4 weeks, then checked again complete blood count, serum fe and serum ferritin. The research results are recorded in a research form and the data is grouped and SPSS version 21.0 software is used for data analysis. A P value <0.05 was considered for statistical analysis. This study was approved by the ethics and research committee of the faculty of medicine, at Hasanuddin University

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Children's Iron deficiency anemia
2. Must be able to drink syrups

Exclusion Criteria:

1. Patients who have diarrhea
2. Patients who experience vomiting
3. Severe anemia
4. Post Transfusion

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
This study was to compare the effect of standard therapy with standard therapy plus vitamin D in children with IDA. | After 4 weeks
  1. Comparing pre-treatment routine blood test, serum iron, and serum ferritin levels between iron supplementation and iron and vitamin D supplementation groups.
  2. Comparing the levels of routine blood tests, serum iron, and serum ferritin results after treatment between iron supplementation and iron and vitamin D supplementation groups.

SECONDARY OUTCOMES:
Comparison of mean changes in complete blood count, serum iron, and serum ferritin level | after 4 weeks
  1. Comparing the difference in routine blood test results, and ferritin before and after treatment between the iron supplementation group and the iron and vitamin D supplementation group.
  2. Comparing the difference of routine blood test results, and serum iron ferritin before and after therapy in the iron supplementation group.
  3. Comparing the difference of routine blood test results, serum iron ferritin before and after therapy in iron supplementation and Vitamin D supplementation groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nadirah R. Ridha, Dr, Study Chair — Hasanuddin University
Locations (1):
- Universitas Hasanuddin, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Samson KLI, Fischer JAJ, Roche ML. Iron Status, Anemia, and Iron Interventions and Their Associations with Cognitive and Academic Performance in Adolescents: A Systematic Review. Nutrients. 2022 Jan 5;14(1):224. doi: 10.3390/nu14010224. PMID 35011099
- See also: The effect of vitamin D supplementation on hemoglobin concentration: a systematic review and meta-analysis — https://nutritionj.biomedcentral.com/articles/10.1186/s12937-020-0526-3
- See also: The effect of iron on vitamin D level in children with combined iron and vitamin D deficiency — https://www.jparathyroid.com/Article/JPD_20180820090934